CLINICAL TRIAL: NCT02529657
Title: Analysis of Effect of Low Level Laser Therapy in Spinal Surgery
Brief Title: Low Level Laser Therapy to Reduce Comorbidity in Spinal Surgery
Acronym: LASPINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Vanessa Milanesi Holanda, MD, MS, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12288113.1.0000.5511
Record Dates: First submitted 2013-11-22; First posted 2015-08-20 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Failed Back Surgery Syndrome
Keywords: Lower Level Laser Therapy (LLLT); inflammation; cytokines; wound healing; laminectomy; clinical study
MeSH Terms: conditions — Failed Back Surgery Syndrome; Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 23 patients were induced to think they will be getting the same treatment, although the LLLT is not operating.
  Interventions: Procedure: Placebo
- Low level Laser Therapy (Experimental): 25 patients were submitted to spine surgery and have received low level laser therapy during surgery, 24 hours after surgery and 48 hours after surgery.
  Interventions: Radiation: Low Level Laser Therapy

INTERVENTIONS:
Radiation: Low Level Laser Therapy — In 23 randomized patients, LLLT (B-Cure, Good Energies ®, Israel), with CW diode laser - semiconductor Gallium Arsenide and aluminum (GaAlAs) will be applied during surgery (λ = 804 nm ± 2 , total exposure time of 240 s, energy density of 2.48 J/cm2 , average power of 40 mW , spot area of 3,876 cm2), in contact mode, for 60 seconds on the laminectomy site, 60 seconds and 120 seconds in the subcutaneous tissue of the skin over the wound bed, respectively. In the first and second day post surgery, will be collected the drainage output for analysis of interleukin 1, 4, 6, 8 and 10 (IL- 1, IL-4, IL -6, IL-8 and IL -10 ) and tumor necrosis factor alpha ( TNF -alpha ).
  Arms: Low level Laser Therapy
Procedure: Placebo — In the operating room, lumbar laminectomy will be performed in 46 patients. During the surgery, 24 hours and 48 hours after surgery, the patients received the regular treatment after laminectomy and were induced to thing that were receiving low level laser therapy in their wound.
  Arms: Placebo

SUMMARY:
Each year, more than one million individuals worldwide are submitted to laminectomies, with a failure rate higher than 40%. Postlaminectomy epidural adhesion is implicated as a main cause of ''failed back surgery syndrome'' and associated with increased risk of complications during revision surgery. The postoperative epidural scar can cause extradural compression or dural tethering, which results in recurrent radicular pain and physical impairment. Several studies in the literature are signalizing that Low-Level-Laser-Therapy (LLLT) is proven to be an effective tool to assist the inflammatory process and wound healing, as well to prevent infection. Thus, the objectives of this project are to delineate and evaluate the LLLT effects in spinal surgery. A prospective randomized, controlled trial with a total of 48 patients who underwent laminectomy, were divided into 2 groups. In the first group, 25 patients received LLLT during the surgical procedure over dura mater, over subcutaneous and on the skin, as well as 24h and 72h post surgery. In the second group, 23 patients were induced to think they will be getting the same treatment, although the laser is not operating. In those groups, C reactive protein, Lactate Dehydrogenase and Creatine kinase were evaluated in the second and fifth days after surgery, digital temperature will be measured and scores in visual analogue scale will be used, 5 minutes pre and 5 minutes post Laser application. The drainage output was collected in the first three days following surgery in both groups. Interleukins were evaluated in interstitial infiltrate drained in 24h and 48h. The data was evaluated for normality and subjected to appropriate statistical analysis, in order to seek representation, as same as the level of significance of the studied samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing to lumbar laminectomy

Exclusion Criteria:

* Active lumbar cancer
* Infectious disease
* Coagulation disorders
* Dural injury during the surgery

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Immunochemistry to evaluate low level laser therapy anti-inflammatory mechanism 24 hours | 24 hours after surgery
  Interstitial infiltrate obtained of Lumbar Drain collected 24 hours after surgery, interleukins IL-1, IL-4, IL-8, IL-10 and TNF alfa were measured through Immunochemistry, using ELISA.
Immunochemistry to evaluate low level laser therapy mechanism 48 hours after light delivery | 48h after surgery
  Interstitial infiltrate was obtained of Lumbar Drain collected 48 hours after surgery, in this infiltrate interleukins IL-1, IL-4, IL-8, IL10 and TNF alfa were measured through Immunochemistry, using ELISA.

SECONDARY OUTCOMES:
Score in Visual Analogue Scale | 5 minutes pre LLLT
  Patient had to choose between 0 and 10 on the 11 point short pain scale.
Score in Visual Analogue Scale | 5 minutes post LLLT
  Change from baseline in pain on the 11 point short pain scale.

OTHER OUTCOMES:
Temperature of the skin in the healing scar | pre and 1 minute post LLLT
  Verified 1 minute before and 1 minute after LLLT
Values of Creatine Kinase in the blood | pre operative, 24h and 48h postoperative
  Obtained through patient blood.
Values of C reactive protein in the blood | pre operative, 24h and 48h postoperative
  Obtained through patient blood pre operative, 24h and 48h postoperative
Values of Lactate dehydrogenase in the blood | pre operative, 24h and 48h postoperative
  Obtained through patient blood pre operative, 24h and 48h postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Chavantes, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho Universtiy, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Farrokhi MR, Vasei M, Fareghbal S, Farrokhi N. The effect of methylene blue on peridural fibrosis formation after laminectomy in rats: an experimental novel study. Spine J. 2011 Feb;11(2):147-52. doi: 10.1016/j.spinee.2011.01.014. PMID 21296299
- [Background] Yildiz KH, Gezen F, Is M, Cukur S, Dosoglu M. Mitomycin C, 5-fluorouracil, and cyclosporin A prevent epidural fibrosis in an experimental laminectomy model. Eur Spine J. 2007 Sep;16(9):1525-30. doi: 10.1007/s00586-007-0344-8. Epub 2007 Mar 27. PMID 17387523
- [Background] Temiz C, Temiz P, Sayin M, Ucar K. Effect of cepea extract-heparin and allantoin mixture on epidural fibrosis in a rat hemilaminectomy model. Turk Neurosurg. 2009 Oct;19(4):387-92. PMID 19847760
- [Background] Oehmichen M. Vitality and time course of wounds. Forensic Sci Int. 2004 Sep 10;144(2-3):221-31. doi: 10.1016/j.forsciint.2004.04.057. PMID 15364394
- [Background] Shah JM, Omar E, Pai DR, Sood S. Cellular events and biomarkers of wound healing. Indian J Plast Surg. 2012 May;45(2):220-8. doi: 10.4103/0970-0358.101282. PMID 23162220
- [Background] Wang R, Ghahary A, Shen Q, Scott PG, Roy K, Tredget EE. Hypertrophic scar tissues and fibroblasts produce more transforming growth factor-beta1 mRNA and protein than normal skin and cells. Wound Repair Regen. 2000 Mar-Apr;8(2):128-37. doi: 10.1046/j.1524-475x.2000.00128.x. PMID 10810039
- [Background] Lee JH, Lee SH. Clinical effectiveness of percutaneous adhesiolysis using Navicath for the management of chronic pain due to lumbosacral disc herniation. Pain Physician. 2012 May-Jun;15(3):213-21. PMID 22622905
- [Background] Tao H, Fan H. Implantation of amniotic membrane to reduce postlaminectomy epidural adhesions. Eur Spine J. 2009 Aug;18(8):1202-12. doi: 10.1007/s00586-009-1013-x. Epub 2009 Apr 30. PMID 19404691
- [Background] Sobottke R, Schluter-Brust K, Kaulhausen T, Rollinghoff M, Joswig B, Stutzer H, Eysel P, Simons P, Kuchta J. Interspinous implants (X Stop, Wallis, Diam) for the treatment of LSS: is there a correlation between radiological parameters and clinical outcome? Eur Spine J. 2009 Oct;18(10):1494-503. doi: 10.1007/s00586-009-1081-y. Epub 2009 Jun 27. PMID 19562386
- [Background] Sandoval MA, Hernandez-Vaquero D. Preventing peridural fibrosis with nonsteroidal anti-inflammatory drugs. Eur Spine J. 2008 Mar;17(3):451-455. doi: 10.1007/s00586-007-0580-y. Epub 2008 Jan 3. PMID 18172695
- [Background] Rochkind S, Drory V, Alon M, Nissan M, Ouaknine GE. Laser phototherapy (780 nm), a new modality in treatment of long-term incomplete peripheral nerve injury: a randomized double-blind placebo-controlled study. Photomed Laser Surg. 2007 Oct;25(5):436-42. doi: 10.1089/pho.2007.2093. PMID 17975958
- [Background] Bae CS, Lim SC, Kim KY, Song CH, Pak S, Kim SG, Jang CH. Effect of Ga-as laser on the regeneration of injured sciatic nerves in the rat. In Vivo. 2004 Jul-Aug;18(4):489-95. PMID 15369190
- [Background] Keskin F, Esen H. Comparison of the effects of an adhesion barrier and chitin on experimental epidural fibrosis. Turk Neurosurg. 2010 Oct;20(4):457-63. doi: 10.5137/1019-5149.JTN.3205-10.2. PMID 20963694
- [Background] LaRocca H, Macnab I. The laminectomy membrane. Studies in its evolution, characteristics, effects and prophylaxis in dogs. J Bone Joint Surg Br. 1974 Aug;56B(3):545-50. No abstract available. PMID 4421702
- See also: Related Info — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisa.jsf